CLINICAL TRIAL: NCT06845228
Title: Kinematic Analysis of Latissimus Dorsi Transfer Results for Shoulder External Rotation Resuscitation with or Without Release of the Subscapularis, in Patients with Neonatal Brachial Plexus Palsy
Brief Title: Kinematic Analysis of Latissimus Dorsi Transfer Results for Shoulder External Rotation Resuscitation
Acronym: CinéLDSS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231773
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Osbtetric Brachial Plexus Palsy
Keywords: Osbtetric Brachial Plexus Palsy; cinematic; latissimus dorsi; infraspinatus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Neonatal brachial plexus palsy is a pathology that remains common and one of its sequelae is lack of external rotation of the shoulder. One of the treatments to increase this range of motion is the transfer of the latissimus dorsi tendon to the infraspinatus muscle. The aim of this study is to analyze the long-term three-dimensional kinematic effects of latissimus dorsi transfer with or without subscapularis release on upper limb joints during the five Mallet tasks and their correlation with clinical and MRI parameters.

Predictive factors such as age at the time of the operation, the extent of the damage and the presence of severe preoperative dysplasia, the presence of neosurgery and the age at which this neosurgery was performed will be evaluated.

The main objective is to evaluate the benefit of releasing the subscapularis during latissimus dorsi transfer surgery in patients with neonatal brachial plexus. This evaluation is done through an analysis of the movement of the upper limb in three dimensions. Kinematic data will be compared between patients with subscapularis release, patients without subscapularis release, and an existing database of unaffected arms.

The secondary objective is to study the correlation between kinematic data and factors that may influence results such as age at the time of surgery, extent of plexus damage, presence of severe preoperative dysplasia , the presence of neosurgery and the age at which this neosurgery was performed. The collection will be done during a single movement analysis session, in a dedicated room at Trousseau hospital, for a duration of approximately 1 hour and 30 minutes.

Part of the equipment designed and manufactured by the Ecole Nationale Supérieure d'Arts et Métiers (ENSAM) for these analyzes will be permanently installed in the analysis room. Other equipment will be installed just before the measurement session and put away at the end. The installation of analysis and measurement equipment as well as the acquisition of data during movements are carried out by ENSAM teacher-researchers or students.

The patient is welcomed into the room by a clinician involved in the study and who will participate in the entire session. In particular, he will carry out a rating of the Mallet score at the start of the session, the placement of sensors for movement analysis, palpation of anatomical points and will give the patient instructions for carrying out the movements.

DETAILED DESCRIPTION:
Patients undergoing latissimus dorsi transfer surgery due to a brachial plexus will be summoned to the ENSAM laboratory. Evaluation of upper limb mobility in 3 dimensions using electromagnetic sensors stuck to the skin from the Fastrak group (Polhemus, Colchester, US). Four segments are included in this analysis (trunk, scapula, humerus, forearm) and two joints are considered: scapulathoracic (ST) and glenohumeral (GH). The hardware used from the Fastrack group includes four receivers (defining technical frameworks) and a stylus (used for scanning purposes).

The transmitter is placed just behind the shoulder blade with the subject in a standing position. Two receivers are fixed on rigid supports which are then connected to the forearm using straps. Two other receptors are fixed directly to the skin using double-sided adhesive tape: a first at the level of the sternum and a second on the flat part of the acromial process of the scapula. The fixing is reinforced with adhesive tape above the sensors. The anatomical frameworks are defined for the trunk, humerus and forearm.

The relative positions of the anatomical and technical frames are defined during a static acquisition phase where the anatomical points defining the anatomical frames are digitized using the stylus, the receptors being simultaneously connected to the segments.

Angular kinematic calculations are then carried out using the anatomical frames and sequences described previously. Finally, eight angular movements are studied: Protraction/retraction, Medial/lateral rotation, and Anterior/posterior rotation for the scapulothoracic joint, angular movements of the elevation plane (GHPE) and elevation (GHEle) and internal/external rotation (GHRot) for the glenohumeral joint.

The subject stands with feet a comfortable width apart and the posterior surface of the heel in contact with an L-shaped mark attached to the floor. In the initial position, the upper limbs are placed in the anatomical reference position (arm alongside the body) for all the tasks described below except for the first where the elbow is flexed to 90° with the forearm in a plane sagittal. To mobilize the upper limb in different directions in space, patients are invited to perform the five tasks of the Mallet score:

* First task: external rotation, elbow to the body and flexed to 90°
* Second task: hand to mouth.
* Third task: hand on the back.
* Fourth task: hand to the neck.
* Fifth task: raise the upper limb in the scapular plane. The scapular plane was defined at 40° from the frontal plane. To normalize the movement, a laser is attached to the external part of the arm and the subject is asked to follow with the laser spot a vertical line which crosses the scapular plane and a plane perpendicular to the scapular plane.

The whole procedure will be successively carried out for the pathological and healthy sides of the patient. For a given side, each task will be repeated three times consecutively and the average value obtained from these three trials will be studied.

For these four previous tasks, in the initial position, the upper limbs were placed in the anatomical reference position.

This evaluation is standardized: The orthopedic surgeon is responsible for the placement of the sensors. The entire procedure is performed successively for the involved side and the intact side. Each task was repeated three times consecutively and the average value obtained from these three trials is studied.

Description of kinematic calculations:

Four segments are included in this kinematic analysis (trunk, scapula, humerus, forearm). Three joints are considered: scapula-thoracic (ST), Gleno-humeral (GH), elbow. In addition to these joints, the movements of the humerus in relation to the trunk (HT) and of the trunk in relation to a fixed reference are also studied. Kinematic measurements will be carried out using the Fastrak electromagnetic tracking device (Polhemus, Colchester, US).It includes four receivers (defining four technical landmarks) and a stylus (used for palpation purposes). The transmitter is placed just behind the shoulder blade, with the subject in a standing position. Two receivers are fixed on rigid supports which are connected to the forearm using straps and to the arm using an cuff. Two other receptors will be directly attached to the skin using hypoallergenic double-sided adhesive tape: to the sternum and to the scapula on the flat part of the acromial process. The fixation is reinforced by hypoallergenic adhesive tape above the sensors. Anatomical landmarks are defined for the trunk, scapula, humerus, and forearm as previously described in Maurel et al., 2013 and Herisson et al. 2017.

The relative positions of the anatomical and technical landmarks are defined during a static acquisition phase where the anatomical points defining the anatomical landmarks are digitized using the stylus, the receptors being simultaneously connected to the segments. The angular kinematic calculations are then carried out using the anatomical landmarks and the sequences described previously (Maurel et al., 2013, Herisson et al. 2017, Maurel et al. 2021) and make it possible to obtain the following angular positions:

* For the scapulothoracic joint: protraction/retraction (STPro), medial/lateral rotation (STMed) and anterior/posterior inclination (STTilt)
* For the glenohumeral joint: elevation plane (GHPE), elevation (GHEle) and internal/external rotation (GHRot)
* For the elbow: flexion/extension and pronation/supination.
* For the movement of the humerus in relation to the trunk: flexion-extension (HTFE), abduction/adduction (HTAbAd) and internal/external rotation (HTRot).
* For the trunk in relation to the fixed reference: flexion-extension (TFE), Inclination (TInc) and axial rotation (TRot).

Software already developed by ENSAM will be used for the kinematic calculations described above, making it possible to obtain the initial and final positions and the amplitudes of each of the angles studied.

The secondary endpoint will focus on the search for correlations between the kinematics of the upper limb previously described and factors that may influence the results such as age at the time of the intervention, the presence of neosurgery and the age at which was performed this neosurgery, the extent of the plexus damage and the presence of severe preoperative dysplasia..

MRIs of the affected shoulder are carried out for the usual follow-up of patients with neonatal brachial plexus damage. The last MRIs carried out after the operation will be analyzed in order to determine morphological parameters such as the glenoid version, the type of glenoid deformity , the percentage of anterior coverage of the humeral head, the shape of the head of the humerus;

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 and 18 years old
* Patients with neonatal brachial plexus
* Patients who had a latissimus dorsi transfer at least two years ago
* Patients with post-operative MRI
* Patients or legal representatives for minors having been informed of the study and having given their informed consent by collection of non-opposition

Exclusion Criteria:

* Legal representatives of minor children or patients who do not understand verbal or written explanations in French
* Patients with bilateral brachial plexus injury

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: University hospital patients aged 6 to 18 with obstetrical brachial plexus injuries
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mallet Score | Through study completion (2 years and 6 month)
  The five tasks of the Mallet score:
  * First task: external rotation, elbow to the body and flexed to 90°
  * Second task: hand to mouth.
  * Third task: hand on the back.
  * Fourth task: hand to the neck.
  * Fifth task: raise the upper limb in the scapular plane. The scapular plane was defined at 40° from the frontal plane. To normalize the movement, a laser is attached to the external part of the arm and the subject is asked to follow with the laser spot a vertical line which crosses the scapular plane and a plane perpendicular to the scapular plane.
  The whole procedure will be successively carried out for the pathological and healthy sides of the patient. For a given side, each task will be repeated three times consecutively and the average value obtained from these three trials will be studied

SECONDARY OUTCOMES:
Confounding factors | Through study completion (2 years and 6 month)
  Study the correlation between kinematic data and factors that may influence results such as age at the time of surgery, extent of plexus damage, presence of severe preoperative dysplasia, presence of neosurgery and the age at which this neosurgery was performed

CONTACTS AND LOCATIONS:
Overall Officials: Franck Fitoussi, PUPH MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Name Service de Chirurgie orthopédique de l'hopital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided